CLINICAL TRIAL: NCT00897299
Title: Identifying Genomic Predictors of Recurrence After Adjuvant Chemotherapy
Brief Title: Identifying Genes That Predict Recurrence in Women With Breast Cancer Treated With Chemotherapy
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000456426; ECOG-E21971CSC; NCI-7613; SANOFI-AVENTIS-ECOG-E21971CSC; GENOMIC-ECOG-E21971CSC
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Estrogen Receptor; Her-2; Pgr
Keywords: estrogen receptor; HER-2; PgR; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict whether cancer will come back after treatment.

PURPOSE: This laboratory study is identifying genes that may help predict recurrence in women with breast cancer treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the prognostic utility of the Oncotype DX™ 21 gene profile for risk of relapse in women with node positive or high-risk node negative breast cancer.
* Identify individual genes whose RNA expression is associated with an increased risk of relapse in these patients.
* Perform an exploratory analysis of individual genes whose RNA expression is associated with an increased risk of relapse differentially in patients previously treated with docetaxel.

OUTLINE: This is a multicenter study.

Tissue samples are examined for association of RNA expression and clinical factors (e.g., tumor size, nodal status, hormone receptor status, age, menopause status), as well as estrogen receptor, progesterone receptor, and HER-2/neu expression by immunohistochemistry and other studies.

PROJECTED ACCRUAL: A total of 900 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Node positive OR high-risk node negative disease
  * Tumor > 1.0 cm in diameter
* No locally advanced, inflammatory, or metastatic breast cancer
* Previously treated with 4 courses of anthracycline-containing chemotherapy (i.e., doxorubicin and docetaxel OR doxorubicin and cyclophosphamide)
* Enrolled on clinical trial ECOG-E2197
* Adequate tumor material available in ECOG Pathology Coordination Center
* Previously consented to future cancer-related research
* Hormone receptor status known

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2005-10-07 (Actual); Primary Completion 2005-10-08 (Actual); Study Completion 2005-10-08 (Actual)

PRIMARY OUTCOMES:
Distant, local/regional, and ipsilateral breast relapse
First breast cancer recurrence
Relapse-free interval

SECONDARY OUTCOMES:
Distant involvement at time of first recurrence
Disease-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Sparano, MD, Study Chair — Albert Einstein College of Medicine; Lori J. Goldstein, MD — Fox Chase Cancer Center

REFERENCES:
- [Result] Badve SS, Baehner FL, Gray R, et al.: ER and PR assessment in ECOG 2197: comparison of locally determined IHC with centrally determined IHC and quantitative RT-PCR. [Abstract] American Society of Clinical Oncology 2007 Breast Cancer Symposium, 7-8 September 2007, San Francisco, California A-87, 2007.
- [Result] Sparano JA, Goldstein L, Childs B, et al.: Association of individual genes with risk of relapse in operable breast cancer: analysis of E2197. [Abstract] American Society of Clinical Oncology 2007 Breast Cancer Symposium, 7-8 September 2007, San Francisco, California A-27, 2007.